CLINICAL TRIAL: NCT05332314
Title: NSAIDs and Time to Union in Diaphyseal Tibia Fractures: Do NSAIDs Make a Difference
Brief Title: NSAIDS vs Opioids in Tibial Fractures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Rodolfo Zamora, MD, Associate Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19.0676
Record Dates: First submitted 2022-04-08; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Anti-Inflammatory Agents, Non-Steroidal; Ibuprofen

STUDY DESIGN:
Intervention Model Description: The study will be a prospective interventional study with two randomized parallel groups.
  Randomization will take place immediately following the identification of a potential participant. The control group will receive the standard of care for diaphyseal tibia fractures. The standard of care consists of intramedullary nailing and post-operative opioids for pain control. The interventional group will have the same surgical indication and intervention but will differ in the primary method of pain control. The study group will receive NSAIDs and a reduced dosage of opioids for pain control. Primary outcome measures will be time to union, non-union, and pain over the post-operative period measured by a VAS pain scale. Once the data collection of both groups is complete, the statistical analysis will begin to determine if there is a statistical difference between the control and study groups in the primary outcome measurements
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NSAIDs (Experimental): This arm is given NSAIDs perioperatively and after discharge
  Interventions: Drug: NSAIDs
- Opioids (No Intervention): This arm will be given the standard opioids treatment to control pain perioperatively and at discharge.

INTERVENTIONS:
Drug: NSAIDs — The patients will be given NSAIDs with a reduced dose of the standard opioids treatment.
  Other Names: Ibuprofen
  Arms: NSAIDs

SUMMARY:
This study will attempt to determine if there is a statistic difference between the time to union, non-union rate and post-operative pain of patients who receive opioids for pain control vs. patients who receive NSAIDs and a reduced dosage of opioids for pain management

DETAILED DESCRIPTION:
The study will be a prospective interventional study with two randomized parallel groups.

Randomization will take place immediately following the identification of a potential participant. The control group will receive the standard of care for diaphyseal tibia fractures. The standard of care consists of intramedullary nailing and post-operative opioids for pain control. The interventional group will have the same surgical indication and intervention but will differ in the primary method of pain control. The study group will receive NSAIDs and a reduced dosage of opioids for pain control. Primary outcome measures will be time to union, non-union, and pain over the post-operative period measured by a VAS pain scale. Once the data collection of both groups is complete, the statistical analysis will begin to determine if there is a statistical difference between the control and study groups in the primary outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 105
* Diaphyseal tibia fracture (OTA/AO 42 A, B)

Exclusion Criteria:

-Tibial fractures not treated with intramedullary nails

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Time to union | through study completion, an average of 1 year
  The time from surgery to bone healing

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Zamora, MD, Principal Investigator — University of Louisville
Locations (2):
- United States (2):
  - University of Louisville Hospital, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giannoudis PV, Hak D, Sanders D, Donohoe E, Tosounidis T, Bahney C. Inflammation, Bone Healing, and Anti-Inflammatory Drugs: An Update. J Orthop Trauma. 2015 Dec;29 Suppl 12:S6-9. doi: 10.1097/BOT.0000000000000465. PMID 26584270
- [Background] Lu C, Xing Z, Wang X, Mao J, Marcucio RS, Miclau T. Anti-inflammatory treatment increases angiogenesis during early fracture healing. Arch Orthop Trauma Surg. 2012 Aug;132(8):1205-13. doi: 10.1007/s00402-012-1525-4. Epub 2012 May 24. PMID 22622792
- [Background] Sathyendra V, Darowish M. Basic science of bone healing. Hand Clin. 2013 Nov;29(4):473-81. doi: 10.1016/j.hcl.2013.08.002. Epub 2013 Oct 15. PMID 24209946
- [Background] Schindeler A, McDonald MM, Bokko P, Little DG. Bone remodeling during fracture repair: The cellular picture. Semin Cell Dev Biol. 2008 Oct;19(5):459-66. doi: 10.1016/j.semcdb.2008.07.004. Epub 2008 Jul 25. PMID 18692584
- [Background] Geusens P, Emans PJ, de Jong JJ, van den Bergh J. NSAIDs and fracture healing. Curr Opin Rheumatol. 2013 Jul;25(4):524-31. doi: 10.1097/BOR.0b013e32836200b8. PMID 23680778
- [Background] Marquez-Lara A, Hutchinson ID, Nunez F Jr, Smith TL, Miller AN. Nonsteroidal Anti-Inflammatory Drugs and Bone-Healing: A Systematic Review of Research Quality. JBJS Rev. 2016 Mar 15;4(3):e4. doi: 10.2106/JBJS.RVW.O.00055. PMID 27500434